CLINICAL TRIAL: NCT03131492
Title: Procalcitonin and C-Reactive Protein as Early Anastomotic Dehiscence Markers in Ovarian Cancer Surgery
Brief Title: Early Dehiscence Markers in Ovarian Cancer Surgery
Acronym: EDMOCS
Status: Completed | Type: Observational
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PR(AMI)68/2017
Record Dates: First submitted 2017-03-24; First posted 2017-04-27 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Ovarian Neoplasms Malignant; Anastomotic Leak
MeSH Terms: conditions — Anastomotic Leak | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Blood test — C-reactive protein and PCT measured preoperatively, and on the second, fourth and sixth postoperative days.

SUMMARY:
EDMOCS trial pretends to evaluate if C-reactive protein (CRP) and procalcitonin (PCT) can predict intestinal anastomotic leaks before early discharge in advanced ovarian cancer surgery requiring intestinal resection. These markers have already been positively tested in colorectal cancer surgery, but not yet in ovarian surgery.

Patients undergoing intestinal resection in ovarian cancer surgery will be included. C-reactive protein and PCT will be measured pre-operatively, and on the second, fourth and sixth postoperative day. Thirty-day readmissions, re-operations and mortality will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Ovarian cancer stage III-IV
* Intestinal resection needed

Exclusion Criteria:

* Infection diagnosed at time of surgery.
* Urgent surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed of an advenced ovarian cancer who need an intestinal resection during ovarian surgery.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Number of patients with anastomotic leak detected by elevation of C-reactive protein and procalcitonin levels | Within the first 30 days after the surgery
  To evaluate whether C-reactive protein (CRP) and procalcitonin (PCT) can predict anastomotic leak before early discharge.

SECONDARY OUTCOMES:
C-reactive protein and procalcitonin measures in patients without complications in ovarian surgery. | Within the first six days after the surgery
  Defining normal range values of C-Reactive Protein and Procalcitonin during postoperative ovarian cancer surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Gil-Moreno, MD, Study Director — Head of Department of Obstetrics and Gynecology, Vall d'Hebron University Hospital; Asunción Pérez-Benavente, MD, Study Director — Head of Unit of Gynecology Oncology Department of Obstetrics and Gynecology; José Luis Sánchez-Iglesias, MD, Principal Investigator — Department of Obstetrics and Gynecology
Locations (1):
- Hospital Universitari de la Vall d'Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Trencheva K, Morrissey KP, Wells M, Mancuso CA, Lee SW, Sonoda T, Michelassi F, Charlson ME, Milsom JW. Identifying important predictors for anastomotic leak after colon and rectal resection: prospective study on 616 patients. Ann Surg. 2013 Jan;257(1):108-13. doi: 10.1097/SLA.0b013e318262a6cd. PMID 22968068
- [Background] Almeida AB, Faria G, Moreira H, Pinto-de-Sousa J, Correia-da-Silva P, Maia JC. Elevated serum C-reactive protein as a predictive factor for anastomotic leakage in colorectal surgery. Int J Surg. 2012;10(2):87-91. doi: 10.1016/j.ijsu.2011.12.006. Epub 2011 Dec 28. PMID 22222182
- [Background] Lu Y, Huang S, Li P, Chen B, Liu W, Chen Z, Yin F. Prognostic evaluation of preoperative serum C-reactive protein concentration in patients with epithelial ovarian cancer. Exp Ther Med. 2015 May;9(5):2003-2007. doi: 10.3892/etm.2015.2350. Epub 2015 Mar 12. PMID 26136929
- [Background] Garcia-Granero A, Frasson M, Flor-Lorente B, Blanco F, Puga R, Carratala A, Garcia-Granero E. Procalcitonin and C-reactive protein as early predictors of anastomotic leak in colorectal surgery: a prospective observational study. Dis Colon Rectum. 2013 Apr;56(4):475-83. doi: 10.1097/DCR.0b013e31826ce825. PMID 23478615
- [Background] Zawadzki M, Czarnecki R, Rzaca M, Obuszko Z, Velchuru VR, Witkiewicz W. C-reactive protein and procalcitonin predict anastomotic leaks following colorectal cancer resections - a prospective study. Wideochir Inne Tech Maloinwazyjne. 2016 Jan;10(4):567-73. doi: 10.5114/wiitm.2015.56999. Epub 2016 Jan 12. PMID 26865894